CLINICAL TRIAL: NCT01096381
Title: A Prospective Clinical Trial Evaluating Potential Biomarkers for Bevacizumab Induced Hypertension
Brief Title: Potential Biomarkers for Bevacizumab-Induced High Blood Pressure in Patients With Solid Tumor
Status: Terminated | Type: Observational
Why Stopped: funding withdrawn due to fellow's departure from VICC
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ingrid Mayer, MD, Assistant Professor of Medicine; Clinical Director, Breast Cancer Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC BRE 0983; P30CA068485 (NIH); VU-VICC-BRE-0983
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer; Cardiovascular Complications; Colorectal Cancer; Fallopian Tube Cancer; Head and Neck Cancer; Lung Cancer; Ovarian Cancer; Peritoneal Cavity Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: cardiovascular complications; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; unspecified adult solid tumor, protocol specific; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; recurrent basal cell carcinoma of the lip; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV squamous cell carcinoma of the lip and oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer; peritoneal cavity cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Fallopian Tube Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Will receive bevacizumab
  Interventions: Other: laboratory biomarker analysis; Other: questionnaire administration
- Will not receive bevacizumab
  Interventions: Other: laboratory biomarker analysis; Other: questionnaire administration

INTERVENTIONS:
Other: laboratory biomarker analysis — Blood collection
Other: questionnaire administration — Survey regarding baseline health and activity level.

SUMMARY:
RATIONALE: Studying samples of blood and urine in the laboratory from patients with cancer receiving bevacizumab may help doctors learn more about changes that occur in DNA and identify biomarkers related to high blood pressure.

PURPOSE: This phase I trial is studying potential biomarkers for bevacizumab-induced high blood pressure in patients with malignant solid tumors, including breast cancer, colorectal cancer, non-small cell lung cancer, head and neck cancer, ovarian cancer, fallopian tube cancer, or primary peritoneal carcinoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To measure the endothelial function over time, including non-invasive assessment of digital-pulse amplitude via Endo-pat test, serum tPA, PAI-1, VEGF, urine TXa2, and PGI-M, in patients with solid malignancies treated with chemotherapy with or without bevacizumab.
* To compare endothelial function changes between patients who develop hypertension (HTN) versus patients who do not develop HTN.

Secondary

* To compare circulating soluble cytokines, proangiogenic factors, glucose tolerance, and cardiac biomarkers over time in these patients.
* To compare endothelial progenitor cell levels pre- and post-bevacizumab in these patients.
* To assess whether physical fitness level at baseline and at 3 months after treatment initiation (assessed subjectively by questionnaire) correlates with relative risk of developing NCI grade ≥ I cardiotoxicity.

OUTLINE: Patients undergo 24-hour blood pressure monitoring at baseline, before second bevacizumab therapy, and periodically during study. Patients also undergo a digital-pulse amplitude measurement periodically during study.

Blood samples are collected at baseline and periodically during study for circulating soluble cytokines, proangiogenic factors, glucose tolerance, cardiac biomarkers, and endothelial progenitor cell level studies. Patients also undergo 24-hour urine sample collection at baseline and periodically during study for protein, creatinine, and metabolites of prostacyclin and thromboxane.

Patients complete physical activity questionnaires at baseline and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

Patients with stage IV or unresectable recurrent cancer (except for renal cell carcinoma and glioblastoma multiforme) that will get bevacizumab as a standard of care, as well as patients about to initiate bevacizumab within the protocols:

* ECOG5103: A Double-Blind Phase III Trial of Doxorubicin and Cyclophosphamide followed by Paclitaxel with Bevacizumab or Placebo in Patients with Lymph Node Positive and High Risk Lymph Node Negative Breast Cancer.
* ECOG1505: A Phase III Randomized Trial of Adjuvant Chemotherapy With or Without Bevacizumab for Patients With Completely Resected Stage IB (> 4 cm) - IIIA Non-Small Cell Lung Cancer (NSCLC)
* ECOG5202: A Randomized Phase III Study Comparing 5-FU, Leucovorin and Oxaliplatin versus 5-FU, Leucovorin, Oxaliplatin and Bevacizumab in Patients with Stage II Colon Cancer at High Risk for Recurrence to Determine Prospectively the Prognostic Value of Molecular Markers
* ECOG1305: Phase III Randomized Trial of Chemotherapy With or Without Bevacizumab in Patients with Recurrent or Metastatic Head and Neck Cancer
* GOG0252: A Phase III Clinical Trial of Bevacizumab With IV Versus IP Chemotherapy in Ovarian, Fallopian Tube and Primary Peritoneal Carcinoma
* GOG0086P: A Three Arm Randomized Phase II Study of Paclitaxel/Carboplatin/Bevacizumab, Paclitaxel/Carboplatin/Temsirolimus, and Ixabepilone/Carboplatin/Bevacizumab as Initial Therapy for Measurable Stage III or IVA, Stage IVB, or Recurrent Endometrial Cancer (Only those arms including bevacizumab)
* GOG0250: A Randomized Phase III Evaluation of Docetaxel and Gemcitabine Plus G-CSF with Bevacizumab Versus Docetaxel and Gemcitabine Plus G-CSF with Placebo in the Treatment of Recurrent or Advanced Leiomyosarcoma of the Uterus
* GOG0240: A Randomized Phase III Evaluation of Docetaxel and Gemcitabine Plus G-CSF with Bevacizumab Versus Docetaxel and Gemcitabine Plus G-CSF with Placebo in the Treatment of Recurrent or Advanced Leiomyosarcoma of the Uterus
* THO0640: A Phase II Multi Center Study Investigating Translational Science in Chemotherapy-Naïve Patients with Stage IIIB or IV Non-Small Cell Lung Cancer (NSCLC) treated with the EGFR-TKI, Erlotinib (SPECS)

Eligibility Criteria:

* Patients ≥ 18 years of age with stage IV or unresectable recurrent cancer (except for renal cell carcinoma and glioblastoma multiforme) that will get bevacizumab as a standard of care.
* Patients ≥ 18 years of age with histologically confirmed breast, colorectal or non-small cell lung (NSCL) cancer that have completed surgical treatment for stages I - III cancer and are going to initiate adjuvant therapy within one of the 3 clinical trials addressing the role of bevacizumab added to chemotherapy in the adjuvant setting of breast, colorectal and NSCL cancer (E5103, E1505 and E5202)
* Patients ≥ 18 years of age with histologically confirmed squamous cell carcinoma of the head and neck (recurrent or metastatic) who are about to initiate chemotherapy with or without bevacizumab within E1305 clinical trial.
* Patients ≥ 18 years of age who are about to initiate chemotherapy with bevacizumab within the following trials: GOG0252, GOG0086P (only those patients receiving bevacizumab arms), GOG0250, and GOG0240.
* Patients ≥ 18 years of age with a histologic diagnosis of non small cell lung cancer who are about to initiate bevacizumab within THO0640 clinical trial.
* Patients must provide informed written consent.

Ineligibility Criteria

- Patients with active renal cell carcinoma or glioblastoma multiforme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage IV breast, colorectal, or non-small cell lung cancer (NSCLC) who will get bevacizumab as a standard of care, as well as patients with breast, colorectal, ovarian/fallopian tube/peritoneal, head and neck, or NSCLC cancer about to initiate bevacizumab. Where possible, the study population will include a control group not receiving bevacizumab.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Digital-pulse amplitude (DPA) measures | 1, 3 and 6 months after initiation of bevacizumab

SECONDARY OUTCOMES:
Relationship between hypertension and baseline DPA | 1, 3 and 6 months
Endothelial progenitor cell levels pre- and post-bevacizumab | 1, 3 and 6 months
Correlation between physical fitness level and cardiotoxicity | 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Mayer, M.D., Principal Investigator — Vanderbilt-Ingram Cancer Center; Ingrid Mayer, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee